CLINICAL TRIAL: NCT04333277
Title: Double-blind Placebo-controlled Clinical Trial of Lactobacillus Helveticus as an add-on Strategy for the Treatment of Major Depression
Brief Title: Lactobacillus Helveticus in the Treatment of Major Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Antonio L Teixeira Jr, Principal Investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE 83541717.0.0000.5149
Record Dates: First submitted 2020-03-25; First posted 2020-04-03 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2020-04

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Patients with major depression (both sexes) will receive capsules with 1 × 10^9 CFUs of Lactobacillus helveticus in addition to a conventional antidepressant treatment for 8 weeks.
  Interventions: Other: Probiotic
- Maltodextrin (Placebo Comparator): Patients with major depression (both sexes) will receive capsules of placebo (maltodextrin) in addition to a conventional antidepressant treatment for 8 weeks
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: Probiotic — Patients with major depression (both sexes) will receive capsules with 1 × 10^9 CFUs of Lactobacillus helveticus in addition to a conventional antidepressant treatment for 8 weeks.
  Arms: Probiotic
Other: Maltodextrin — Patients with major depression (both sexes) will receive capsules of placebo (maltodextrin) in addition to a conventional antidepressant treatment for 8 weeks
  Arms: Maltodextrin

SUMMARY:
The main objective of the study is to evaluate whether the association of the probiotic Lactobacillus helveticus to standard antidepressant will contribute to the treatment of major depression.

DETAILED DESCRIPTION:
Patients with the diagnosis of major depression according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria will receive one daily oral dose of 1 × 10^9 colony-forming units (CFUs) of Lactobacillus helveticus or placebo for 8 weeks in addition to conventional antidepressant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years old;
* Diagnosis of major depression
* Agree to sign the informed consent.

Exclusion Criteria:

* Treatment with anti-inflammatory drugs or antibiotics of any pharmacological classes in the month before treatment enrollment;
* Use of dietary supplementation (herbal supplements, other pro- or prebiotics).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Change in the depressive symptoms severity | 8 weeks
  Depression symptoms severity will be assessed through the Montgomery-Asberg Depression Rating Scale (MADRS) (Minimum: 0 to 6 - normal/symptom absent/ Maximum: >34 - severe depression). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in microbiota composition | 8 weeks
  Microbiota composition will be assessed by Real-Time qPCR.
Changes in the serum levels of biomarkers | 8 weeks
  Inflammatory markers (adiponectin, resistin, leptin, TNF, IL6 and IL10) and neurotrophic factors (GDNF, NGF) will be assessed by enzyme-linked immunosorbent assay (ELISA). Markers will be measured in pg/ml.
Change in perception of stress | 8 weeks
  Perception of stress will be assessed by Perceived Stress Scale (PSS). It is a measure of the degree to which life situations are assessed as stressful. Range from 0 to 40 with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Aline Silva de Miranda, PhD, Study Chair — Federal University of Minas Gerais; Érica Leandro Marciano Vieira, Study Chair — Federal University of Minas Gerais; Lais Bhering Martins, Study Chair — Federal University of Minas Gerais
Locations (1):
- Hospital das Clínicas, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided